CLINICAL TRIAL: NCT05675241
Title: Characterizing the Inflammation Around Dental Implants: Bacterial Infection, Hypersensitivity, or Both?
Brief Title: Characterizing the Inflammation Around Dental Implants
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: McGill University (Other)
Collaborators: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-7639
Record Dates: First submitted 2022-12-22; First posted 2023-01-09 (Actual); Last update posted 2023-01-09 (Actual); Status verified 2022-12

CONDITIONS: Peri-Implantitis; Peri-implant Mucositis; Implant Site Reaction; Implant Site Infection; Hypersensitivity; Implant Site Rash; Implant Infection
Keywords: Peri-implantitis; Peri-implant Mucositis; Hypersensitivity; Dental Implant Failure; Inflammatory Mediators
MeSH Terms: conditions — Peri-Implantitis; Hypersensitivity | interventions — Diagnostic Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Peri-implant crevicular fluid
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Functional Dental Implant: An implant restored with a prothesis and in function for a minimum of one year.
  Interventions: Diagnostic Test: Clinical examination of a dental implant; Diagnostic Test: Radiological Examination; Diagnostic Test: Peri-implant crevicular fluid sample collection

INTERVENTIONS:
Diagnostic Test: Clinical examination of a dental implant — Clinical examination includes bleeding on probing, pocket depth, gingival biotype, suppuration, gingival index
Diagnostic Test: Radiological Examination — A standardized periapical radiograph in parallax technique will be taken.
Diagnostic Test: Peri-implant crevicular fluid sample collection — A sample of the peri-implant crevicular fluid will be collected using paper strip for 60 seconds. The sample of the fluid will be a resultant of inserting six different strips at the same time in six sites of the implant including mesiobuccal, midbuccal, distobuccal, distopalatal/distolingual, midpalatal/midlingual, mesiopalatal/mesiolingual sites of the implant.

SUMMARY:
The use of titanium dental implants has become a common modern treatment to restore teeth. Although the success rate of dental implants is high, inflammation around the dental implant still occurs. The current study will investigate if the inflammation around the implant is due to bacterial infection, hypersensitivity or both.

The goal of this cross-sectional study is to (1) Establish the levels of cytokines in peri-implant crevicular fluid associated with bacterial infection and hypersensitivity reaction; (2) Compare the levels of cytokines associated with hypersensitivity and bacterial infection between healthy implants and inflamed implants (peri-mucositis and peri-implantitis); (3) Determine whether the difference in the levels of cytokines, if they exist, reflects the clinical diagnosis of healthy implants and inflamed implants.

DETAILED DESCRIPTION:
The main objective of this study is to:

1. Establish the levels of cytokines in peri-implant crevicular fluid associated with bacterial infection (Type 1 and 3: IL-1, IL-6, IL-12, IL-17, IL-23, GM-CSF, IFN-γ, TNF-α), hypersensitivity reaction (Type 2: IL-4, IL-5, and IL-13) and the level of MMPs and including MMP-1, MMP-2, MMP-3, MMP-9 and MMP-13.
2. Compare the levels of cytokines associated with hypersensitivity and bacterial infection between healthy implants and inflamed implants (peri-mucositis and peri-implantitis).
3. Determine whether the difference in the levels of cytokines, if they exist, reflects the clinical diagnosis of healthy implants and inflamed implants.

Secondary objectives includes:

1. Measure the volume of peri-implant crevicular fluid and compare it between healthy implants and inflamed implants (peri-mucositis and peri-implantitis).
2. Investigate the association between the levels of cytokines and the severity of inflammatory responses.
3. Show how levels of cytokines influence the severity of inflammatory responses.

ELIGIBILITY:
Inclusion Criteria:

* Received at least one functional implant (implant restored with a prothesis);
* Did not receive peri-implant mucositis and peri-implantitis treatment in the past three months.

Exclusion criteria:

* Dental records with incomplete information;
* Individuals with a weak immune system or chronic disease such as diabetes, heart, lung or kidney disease;
* Pregnant women;
* Individuals undergoing orthodontic therapy and those who have oral piercing.
* History of diseases that modify or suppress the immune and inflammatory response, including rheumatoid arthritis, diabetes, lupus, and inflammatory bowel disease and metastatic cancer;
* Taking medications that cause antiresorptive osteonecrosis of the jaw (including any dose of intravenous bisphosphonates, oral bisphosphonate intake for more than three years, receptor activator of nuclear factor kappa-B ligand inhibitors, or antiangiogenic medications);
* Taking medications known to induce gingival hyperplasia including anticonvulsants, immunosuppressants, or calcium channel blockers;
* Taking steroid medications, systemic or local antibiotics in the last three months (as this may affect the interleukins activity);
* Received radiation therapy to the head and neck or chemotherapy;
* Received treatment to manage an inflamed implant, including management of peri-implantitis and peri-implant mucositis in the last three months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: This cross-sectional study is carried out at McGill University Health Center (MUHC) - Montreal General Hospital Oral and Maxillofacial Clinic. The electronic dental records database at the MUHC Montreal General Hospital Oral and Maxillofacial clinic were screened to identify potentially eligible participants. Individuals who had a functional implant (implant restored with a prosthesis) placed between year 2010 and year 2016 were reviewed. Eligible individuals are contacted and invited to participate.
Sampling Method: Non-Probability Sample
Enrollment: 177 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Health status of the implant | Baseline (Cross-sectional)
  Classifying the implant into healthy implant, peri-implant mucositis and peri-implantitis according to the 2017 World Workshop (Berglundh et al. 2018).
Levels of inflammatory mediators in Periimplant crevicular fluid | Baseline (Cross-sectional)
  Establishing the the levels of cytokines in peri-implant crevicular fluid associated with bacterial infection (Type 1 and 3: IL-1, IL-6, IL-12, IL-17, IL-23, GM-CSF, IFN-γ, TNF-α), hypersensitivity reaction (Type 2: IL-4, IL-5, and IL-13) and the level of MMPs and including MMP-1, MMP-2, MMP-3, MMP-9 and MMP-13.

SECONDARY OUTCOMES:
Gingival Crevicular fluid volume | Baseline (Cross-sectional)
  Measuring the volume of peri-implant crevicular fluid using Periotron device. The measurement unit is μL.

CONTACTS AND LOCATIONS:
Overall Officials: Heba Allah Madi Dr, Principal Investigator — McGill University; Jocelyne Feine Dr, Study Chair — McGill University; Nicholas Makhoul Dr, Study Director — McGill University & McGill University Health Centre
Locations (1):
- Montreal General Hospital - Oral & Maxillofacial Surgery Clinic, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data (IPD) available to other researchers.

REFERENCES:
- [Background] Berglundh T, Armitage G, Araujo MG, Avila-Ortiz G, Blanco J, Camargo PM, Chen S, Cochran D, Derks J, Figuero E, Hammerle CHF, Heitz-Mayfield LJA, Huynh-Ba G, Iacono V, Koo KT, Lambert F, McCauley L, Quirynen M, Renvert S, Salvi GE, Schwarz F, Tarnow D, Tomasi C, Wang HL, Zitzmann N. Peri-implant diseases and conditions: Consensus report of workgroup 4 of the 2017 World Workshop on the Classification of Periodontal and Peri-Implant Diseases and Conditions. J Clin Periodontol. 2018 Jun;45 Suppl 20:S286-S291. doi: 10.1111/jcpe.12957. PMID 29926491
- [Background] Baseri M, Radmand F, Hamedi R, Yousefi M, Kafil HS. Immunological Aspects of Dental Implant Rejection. Biomed Res Int. 2020 Dec 9;2020:7279509. doi: 10.1155/2020/7279509. eCollection 2020. PMID 33376734
- [Background] Annunziato F, Romagnani C, Romagnani S. The 3 major types of innate and adaptive cell-mediated effector immunity. J Allergy Clin Immunol. 2015 Mar;135(3):626-35. doi: 10.1016/j.jaci.2014.11.001. Epub 2014 Dec 18. PMID 25528359
- [Background] Poli PP, de Miranda FV, Polo TOB, Santiago Junior JF, Lima Neto TJ, Rios BR, Assuncao WG, Ervolino E, Maiorana C, Faverani LP. Titanium Allergy Caused by Dental Implants: A Systematic Literature Review and Case Report. Materials (Basel). 2021 Sep 12;14(18):5239. doi: 10.3390/ma14185239. PMID 34576463
- [Background] Lee CT, Huang YW, Zhu L, Weltman R. Prevalences of peri-implantitis and peri-implant mucositis: systematic review and meta-analysis. J Dent. 2017 Jul;62:1-12. doi: 10.1016/j.jdent.2017.04.011. Epub 2017 May 3. PMID 28478213